CLINICAL TRIAL: NCT01733823
Title: Phase I/II Study on Accelerated, Hyperfractionated Radiotherapy With Concomitant Cisplatin and Nimorazole for Patients With Stage III-IV p16 Negative Squamous Cell Cancer (SCC) of the Larynx, Pharynx and Oral Cavity
Brief Title: DAHANCA 28A: Phase I/II Study on Accelerated, Hyperfractionated Radiotherapy With Concomitant Cisplatin and Nimorazole
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Danish Head and Neck Cancer Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAHANCA 28A
Record Dates: First submitted 2012-11-08; First posted 2012-11-27 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: HNSCC,Larynx, Pharynx and Oral Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Diseases | interventions — Cisplatin; Nimorazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): Performance scale 0-1, Charlson co-morbidity score=0 Treatment: 76 Gy/ 56 fx/ 10/W with cisplatin 40 mg/m2/W and nimorazole
  Interventions: Radiation: 76 Gy/ 56 fx/ 10/W with cisplatin 40 mg/m2/W and nimorazole
- Group B (Experimental): PS 0-1 Charlson=1 Treatment: 76 Gy/ 56 fx/ 10/W with cisplatin 40 mg/m2/W and nimorazole
  Interventions: Radiation: 76 Gy/ 56 fx/ 10/W with cisplatin 40 mg/m2/W and nimorazole
- Group C (Experimental): PS 0-1 Charlson >=2 Will start inclusion after Group A and B Treatment: 76 Gy/ 56 fx/ 10/W with cisplatin 40 mg/m2/W and nimorazole
  Interventions: Radiation: 76 Gy/ 56 fx/ 10/W with cisplatin 40 mg/m2/W and nimorazole
- Group D (Experimental): PS 2, Charlson: Any Will start inclusion after Group C Treatment: 76 Gy/ 56 fx/ 10/W with cisplatin 40 mg/m2/W and nimorazole
  Interventions: Radiation: 76 Gy/ 56 fx/ 10/W with cisplatin 40 mg/m2/W and nimorazole

INTERVENTIONS:
Radiation: 76 Gy/ 56 fx/ 10/W with cisplatin 40 mg/m2/W and nimorazole

SUMMARY:
P16 negative cancers continue to have a dismal prognosis despite advances in the treatment of head and neck cancer. Acceleration, dose-escalation, hyperfractionation, chemotherapy and nimorazole has been shown to improve local control. The purpose of the study i to investigate the level of co-morbidity and performance status (PS) that allows the combination of all of the above means of treatment intensification

ELIGIBILITY:
Inclusion Criteria:

* Squamous Cell Carcinoma head and neck cancer of the pharynx, larynx and oral cavity
* P16 negative
* T1-4
* N1-3
* M0
* Organ function and performance status allowing radical chemo-radiotherapy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Compliance | End of radiotherapy (approximately 5.5 weeks after start of radiotherapy)
  Proportion of patients that receive radiotherapy in accordance to prescribed dose and treatment time

SECONDARY OUTCOMES:
Acute toxicity | 2 months after end of radiotherapy
  In accordance with the Danish Head and Neck Cancer Group (DAHANCA) toxicity scales
Response rate | 2 months after end of radiotherapy
  Proportion of complete and partial responders

CONTACTS AND LOCATIONS:
Overall Officials: Jens Overgaard, MD, DMSc, Principal Investigator — Danish Head and Neck Cancer Group
Locations (4):
- Denmark (4):
  - Aarhus, Aarhus, Aarhus C
  - Odense, Odense, Odense C
  - Aalborg, Aalborg
  - Herlev, Herlev